CLINICAL TRIAL: NCT03226379
Title: Integrating the Diagnosis and Management of HIV-associated Central Nervous System (CNS) Infections Into Routine Health Services in Low and Middle Income Countries (LMICs)
Brief Title: Driving Reduced AIDS-associated Meningo-encephalitis Mortality
Acronym: DREAMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); National Agency for Research on AIDS and Viral Hepatitis (ANRS) (Other); Institut Pasteur (Industry); National Institute for Medical Research, Tanzania (Other Government); Amana Hospital, Dar es Salaam, Tanzania (Unknown); University of North Carolina Project-Malawi (UNC Project), Lilongwe, Malawi (Unknown); Kamuzu Central Hospital (Other); Yaounde Central Hospital (Other Government); Zomba Central Hospital, Zomba, Malawi (Unknown); Lighthouse Trust (Other); Mwananyamala Hospital, Dar es Salaam, Tanzania (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 16.0091
Record Dates: First submitted 2017-05-31; First posted 2017-07-21 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: AIDS-Related Opportunistic Infections; Meningo-encephalitis; Cryptococcal Meningitis; Bacterial Meningitis; Tuberculous Meningitis; Cerebral Toxoplasmosis
Keywords: HIV related Meningitis; AIDS-Related Opportunistic Infections; Advanced HIV Disease; Health Systems Strengthening; Education Programmes
MeSH Terms: conditions — AIDS-Related Opportunistic Infections; Meningitis, Cryptococcal; Meningitis, Bacterial; Tuberculosis, Meningeal; Toxoplasmosis, Cerebral

STUDY DESIGN:
Intervention Model Description: Cohort study with a before and after design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DREAMM (Other): 4 DREAMM interventions to reduce HIV-related meningoencephalitis mortality once access to essential diagnostic tests and medicines:
  1. Health system strengthening
  2. Delivery of a co-designed education program tailored to frontline healthcare workers
  3. Implementation of an algorithm for HIV-related meningoencephalitis
  4. Infectious diseases/AHD mentorship and laboratory capacity building
  Interventions: Other: DREAMM

INTERVENTIONS:
Other: DREAMM — 4 DREAMM interventions to reduce HIV-related meningoencephalitis mortality once access to essential diagnostic tests and medicines:
  1. Health system strengthening
  2. Delivery of a co-designed education program tailored to frontline healthcare workers
  3. Implementation of an algorithm for HIV-related meningoencephalitis
  4. Infectious diseases/AHD mentorship and laboratory capacity building

SUMMARY:
The DREAMM project is investigating whether the DREAMM interventions (1) Health system strengthening, 2) Co-designed education programs tailored to frontline healthcare workers, 3) Implementation of a diagnostic and treatment algorithm and, 4) Communities of practice in infectious diseases and laboratory capacity building) when combined reduce two week all-cause mortality of HIV-associated meningo-encephalitis in African LMICs.

DETAILED DESCRIPTION:
HIV-associated central nervous system (CNS) infection causes significant mortality and places a high burden on limited health care resources in Sub-Saharan Africa (SSA). Cohort and autopsy studies estimate that CNS infections cause up to a third of HIV-related deaths in African LMICs.

Cryptococcal meningitis alone is estimated to account for up to 20% of HIV-related mortality and its' incidence in Africa, unlike in resource-rich settings, has remained high despite antiretroviral roll out.

In African low and middle-income countries (LMICs) mortality associated with cryptococcal meningitis has been estimated at 70% at 3 months.

Tuberculous meningitis mortality also remains unacceptably high and is reported at over 70% in a study from Cameroon. Delays in diagnosis are key causes of poor patient outcomes for tuberculous and bacterial meningitis, and cryptococcal meningitis where patients present late and with advanced disease.

The aim of the DREAMM study is to drive down this unacceptably high mortality associated with HIV-associated meningo-encephalitis in LMICs.

A further aim is to provide capacity building in implementation research at each of the sites driven by the local African Principal Investigators (PIs) (Dr Cecilia Kanyama, Lilongwe, Malawi; Dr Charles Kouanfack, Yaoundé, Cameroon; Dr Sayoki Mfinanga, NIMR, Dar es Salaam Tanzania, Dr Saulos Nyirenda, Zomba, Malawi).

The project is in three phases:

1. Observation: Local clinical and laboratory procedures and practices and availability of essential drugs and diagnostic tests for routine care of HIV-associated meningo-encephalitis patients in three study countries will be observed and documented. 75 patients in total will be recruited into the observation phase of DREAMM, 25 patients from each study country.
2. Training: A co-designed laboratory and clinical training program on HIV-associated meningitis in LMICs tailored to frontline healthcare workers (HCWs) will be delivered. Key clinical and laboratory routine HCWs will be trained including on the latest point of care (POC) diagnostic tests and safe administration of essential medicines for HIV-associated meningo-encephalitis such as amphotericin B deoxycholate using a Train the Trainer approach. The knowledge and skills will be disseminated widely following this training by frontline HCWs. Locally adapted optimal clinical and laboratory pathways for the diagnosis and treatment of HIV-related meningoencephalitis in resource limited settings will be devised during the training phase using a health system engineering approach.
3. Implementation: Implementation of an algorithmic approach to diagnosis and treatment of HIV-associated meningitis including aggressive microbiological detection and treatment of cryptococcosis and tuberculosis in the five study sites. The aim is to reduce the time from participant presentation to diagnostic testing and administration of effective, microbiologically-driven treatment. As part of the implementation of the algorithm, the optimised clinical and laboratory pathways endorsed by local leadership are implemented. Communities of practice are formed with weekly multidisciplinary meetings to discuss clinical cases and continue laboratory capacity building.

The data from the observation and implementation phases of the study will be fed back to local ministries of health (MOH), and access to essential antifungal drugs and diagnostic tests for HIV-associated meningitis improved and finally, cohesive HIV-related meningitis guidelines for African LMICs developed.

Important sub-studies include a health economics evaluation study to determine the cost of the intervention and routine care costs. A new semi-quantitative cryptococcal antigen lateral flow assay (CrAg LFA) (CryptoPS, Biosynex, Strasburg, France) will be evaluated uniquely for the diagnosis of patients with meningo-encephalitis. New, POC polyvalent tests (CrAg/HIV) and (CrAg/Streptococcus pneumoniae) will also be evaluated.

These POC tests nested within algorithms, and the new tests being evaluated, together with administration of recommended, microbiologically driven treatments have the potential to significantly reduce CNS infection-related mortality by reducing delays in proven diagnosis and initiation of effective treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients > 18 years with 1st episode of suspected meningo- encephalitis
2. Known to be HIV positive or willing to undertake an HIV test
3. Willing to agree to participate in the study

Exclusion Criteria:

1. Patients presenting with suspected relapse of HIV-associated meningo-encephalitis
2. HIV negative patients
3. Pregnant or lactating patients
4. Patients presenting with a known diagnosis of primary CNS Lymphoma or cerebral malaria
5. COVID-19 infected patients

Patients who are HIV negative or are diagnosed with cerebral malaria on hospital admission or after initial investigation will be excluded or withdrawn from the DREAMM study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2016-04-23 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
2-week all-cause mortality | 2 weeks from enrolment
  2-week all-cause mortality from enrolment

SECONDARY OUTCOMES:
10-week all-cause mortality | 10 weeks from enrolment
  10-week all-cause mortality from enrolment
4-week all-cause mortality | 4 weeks from enrolment
  4-week all-cause mortality 4 weeks from enrolment
10-week and 6-month rate of death | 10 weeks and 6 months from enrolment
  10-week and 6-month rate of death 10 weeks and 6 months from enrolment
Time to appropriate investigation: lumbar puncture, brain imaging | 10 weeks from enrolment
  Time to appropriate investigation: lumbar puncture, brain imaging 10 weeks from enrolment
Time to appropriate, microbiologically guided treatment | 10 weeks from enrolment
  Time to appropriate, microbiologically guided treatment 10 weeks from enrolment
Prevalence of cryptococcal, tuberculous and bacterial meningitis and toxoplasma meningo-encephalitis and neurosyphilis | 10 weeks from enrolment
  Prevalence of cryptococcal, tuberculous and bacterial meningitis and toxoplasma 10 weeks from enrolment
Time to ART initiation | 10 weeks from enrolment
  Time to ART initiation 10 weeks from enrolment
6-month all-cause mortality | 6 months from enrolment
  6-month all-cause mortality 6 months from enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Angela Loyse, MD, Principal Investigator — St George's, University of London
Locations (5):
- Hôpital Central Yaoundé, Yaoundé, Cameroon
- Malawi (2):
  - Kamuzu Central Hospital, Lilongwe
  - Zomba Central Hospital, Zomba
- Tanzania (2):
  - Amana Hospital, Dar es Salaam
  - Mwananyamala Hospital, Dar es Salaam

REFERENCES:
- [Derived] Mfinanga S, Kanyama C, Kouanfack C, Nyirenda S, Kivuyo SL, Boyer-Chammard T, Phiri S, Ngoma J, Shimwela M, Nkungu D, Fomete LN, Simbauranga R, Chawinga C, Ngakam N, Heller T, Lontsi SS, Aghakishiyeva E, Jalava K, Fuller S, Reid AM, Rajasingham R, Lawrence DS, Hosseinipour MC, Beaumont E, Bradley J, Jaffar S, Lortholary O, Harrison T, Molloy SF, Sturny-Leclere A, Loyse A; DREAMM Consortium. Reduction in mortality from HIV-related CNS infections in routine care in Africa (DREAMM): a before-and-after, implementation study. Lancet HIV. 2023 Oct;10(10):e663-e673. doi: 10.1016/S2352-3018(23)00182-0. PMID 37802567